CLINICAL TRIAL: NCT04715997
Title: A Phase 1/2a, Multicenter, Randomized, Double-blind, Placebo-controlled Study to Investigate the Safety, Tolerability, and Immunogenicity of GX-19N, a COVID-19 Preventive DNA Vaccine in Healthy Subjects
Brief Title: Safety and Immunogenicity Study of GX-19N, a COVID-19 Preventive DNA Vaccine in Healthy Adults
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Genexine, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Prevention
Other Study IDs: GX-19N-HV-002
Record Dates: First submitted 2021-01-18; First posted 2021-01-20 (Actual); Last update posted 2025-08-20 (Actual); Status verified 2022-11

CONDITIONS: SARS-CoV-2
MeSH Terms: interventions — GX-19N vaccine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GX-19: Dose A (Experimental): Dose A of GX-19N will be intramusculary administered via EP on day 1 and day 29.
  Interventions: Drug: GX-19N
- Placebo: Normal saline (Placebo Comparator): Placebo will be intramusculary administered via EP on day 1 and day 29.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: GX-19N — DNA vaccine expressing SARS-CoV-2 S-protein antigen including the Nucleocapsid protein (NP) antigen
  Other Names: Dose A
  Arms: GX-19: Dose A
Drug: Placebo — Normal saline
  Other Names: Normal saline
  Arms: Placebo: Normal saline

SUMMARY:
The objective of our study is to evaluate safety, tolerability, and immunogenicity of COVID-19 preventive DNA vaccine in healthy volunteers.

DETAILED DESCRIPTION:
This clinical study is phase 1/2a clinical trial to evaluate safety, tolerability, and immunogenicity of COVID-19 preventive vaccine by intramuscularly administration in healthy volunteers.

Phase 1 of this study is designed as single arm, open-labeled and a total of 20 subjects will be enrolled. Phase 2a of study is designed as randomized, double-blind, placebo controlled and a total of 150 subjects are planned to be enrolled.

ELIGIBILITY:
Inclusion Criteria:

* Able and willing to comply with all study procedures and voluntarily signs informed consent form
* Healthy adult male or female aged 19-55 years
* Willing to provide specimens such as blood and urine during the study, including end of study visit.

Exclusion Criteria:

* Immunosuppresion including immunodeficiency disease or family history
* Any history of malignant disease within the past 5 years
* Scheduled to undergo any surgery or dental treatment during the study
* Having received immunoglobulin or blood-derived drugs or being expected to be administered within 3 months prior to administration.
* Having relied on antipsychotic drugs and narcotic analgesics within 6 months before administration
* Positive of serology test at screening
* Suspected of drug abuse or a history within 12 months prior to administration
* Active alcohol use or history of alcohol abuse
* Serious adverse reaction to a drug containing GX-19N or other ingredients of the same categories or to a vaccine or antibiotic, nonsteroidal anti-inflammatory disease control, etc. or an allergic history
* History of hypersensitivity to vaccination such as Guillain-Barre syndrome
* Those who have or with a history of disease corresponding to other hepatobiliary, kidneys, nervous systems (middle or peripheral), respiratory machines (e.g. asthma, pneumonia, etc., endocrine systems (uncontrolled diabetes, hyperlipidemia, etc.) and cardiovascular (congestive heart failure, coronary artery disease, myocardial infarction, uncontrolled hypertension), blood tumors, urinary machines, mental, musculoskeletal systems, immune system (rheumatoid arthritis, systemic arthritis, mumps, immunodeficiency disease)
* Having hemophilia at risk of causing serious bleeding when injected intramuscularly or receiving anticoagulants
* Subjects who have been contact with COVID-19 infections in the past prior to administration, have been classified as COVID-19 confirmed patients, medical patients or patients with symptoms or have been identified with SARS and MERS infection history in the past
* Acute fever, cough, difficulty breathing, chills, muscle aches, headache, sore throat, loss of smell, or loss of taste within 72 hours prior to administration
* Other vaccination history within 28 days prior to the administration or being scheduled to be inoculated during the study
* History of having taken immunosuppressant or Immune modifying drug within 3 months prior to administration
* Having participated and had clinical trial drug administration in another clinical trial or biological equivalence study within 6 months prior to the administration
* Pregnant or breastfeeding female, however, those are allowed to participate in the study only if they stop breastfeeding before participation (fertile female† must be negative in serum pregnancy test at screening
* Fertile female who do not agree to use effective contraception methods (condoms, contraceptive diaphragm, intrauterine contraceptive devices) during the study
* Any other clinically significant medical or psychiatric finding which is considered inappropriate by investigator

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 185 (Actual)
Dates: Start 2020-12-30 (Actual); Primary Completion 2022-04-19 (Actual); Study Completion 2022-04-19 (Actual)

PRIMARY OUTCOMES:
Incidence of Solicited Adverse Events | Through 1 year post vaccination
  solicited local and systemic AEs after vaccination
Incidence of Unsolicited Adverse Events | Through 1 year post vaccination
  unsolicited AEs after vaccination
Incidence of Serious Adverse Events | Through 1 year post vaccination
  percentage of subjects with SAEs

SECONDARY OUTCOMES:
GMT of Antigen-specific Binding Antibody Titers | Through 1 year post vaccination
  Geometric mean titer (GMT) of antigen-specific binding antibody after vaccination
GMFR of Antigen-specific Binding Antibody Titers | Through 1 year post vaccination
  Geometric mean fold rise (GMFR) of antigen-specific binding antibody after vaccination
Percentage of Subjects Who Seroconverted After Vaccination | Through 1 year post vaccination
  Seroconversion defines when FRNT50 is detected more than four times from the baseline after vaccination
GMT and GMFR of Neutralizing Antibody Level | Through 1 year post vaccination
  Geometric mean titer (GMT) and Geometric mean fold rise (GMFR) of neutralizing antibody after vaccination
GMFR of Neutralizing Antibody Level | Through 1 year post vaccination
  Geometric mean fold rise (GMFR) of neutralizing antibody after vaccination
GMSN and GMFR of Spot Forming Unit (SFU) detected by IFN-gamma ELISPOT assay | Through 1 year post vaccination
  Geometric mean spot numbers (GMSN) and Geometric mean fold rise (GMFR) of SFU after vaccination

OTHER OUTCOMES:
Change From Baseline in Antigen-specific IFN-gamma Cellular Immune Response | Through 1 year post vaccination
  Antigen-specific IFN-γ T cell immune response assessed after vaccination

CONTACTS AND LOCATIONS:
Overall Officials: JungWon Woo, Ph.D., Study Director — Genexine, Inc.; Jun Yong Choi, MD, Principal Investigator — Severance Hospital
Locations (5):
- South Korea (5):
  - KyungHee University Medical Center, Seoul
  - Severance Hospital, Seoul
  - Hanyang University Hospital, Seoul
  - Gangnam Severance Hospital, Seoul
  - Ajou University Hospital, Suwon

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ahn JY, Lee J, Suh YS, Song YG, Choi YJ, Lee KH, Seo SH, Song M, Oh JW, Kim M, Seo HY, Kwak JE, Youn JW, Woo JW, Shin EC, Sung YC, Park SH, Choi JY. Safety and immunogenicity of two recombinant DNA COVID-19 vaccines containing the coding regions of the spike or spike and nucleocapsid proteins: an interim analysis of two open-label, non-randomised, phase 1 trials in healthy adults. Lancet Microbe. 2022 Mar;3(3):e173-e183. doi: 10.1016/S2666-5247(21)00358-X. Epub 2022 Feb 8. PMID 35156068